CLINICAL TRIAL: NCT06801912
Title: A Behavior Change Technique (BCT) Intervention to Develop an Hourly Activity Habit Among Caregivers for Persons Alzheimer's Disease (AD) or Alzheimer's Disease Related Dementias (ADRD)
Brief Title: A BCT Intervention for an Hourly Activity Habit Among Caregivers for Persons With AD/ADRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-0042; 2P30AG063786 (NIH)
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Sedentary Behavior
Keywords: caregiver; Alzheimer's disease; Alzheimer Related Dementia; behavior change techniques; habit formation; sedentary behavior
MeSH Terms: conditions — Sedentary Behavior; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This will be a 12-week, NIH Stage II Behavioral Trial, consisting of a single-arm, multi-component, personalized BCT intervention trial, enrolling caregivers of persons with AD/ADRD. Participants will be provided with 4 BCTs daily (Goal Setting, Action Planning, Self-Monitoring, and Prompts/Cues) that have been associated with habit formation theory and development of physical activity habits in prior research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavior Change Technique Package (Experimental): This will be a 12-week, single-arm, multi-component, personalized BCT intervention. Participants will be provided with 4 BCTs daily (Goal Setting, Action Planning, Self-Monitoring, and Prompt/Cue) that have been associated with habit formation theory and development of physical activity habits in prior research.
  Interventions: Behavioral: Behavior Change Technique Package

INTERVENTIONS:
Behavioral: Behavior Change Technique Package — Behavior Change Technique 1: Goal setting (Behavior) (BCT 1.1). Goal setting for behavior is defined as setting a goal for the behavior to be achieved.
  Behavior Change Technique 2: Action planning (BCT 1.4). Action planning is defined as detailing the plan of where, for how long, and at what time taking medication is going to be performed.
  Behavior Change Technique 3: Self-monitoring of behavior (BCT 2.3). Self-monitoring of behavior is defined as monitoring and recording behavior.
  Behavior Change Technique 4: Prompts/Cues (BCT 7.1) This BCT is defined as prompt rehearsal and repetition of the behavior in the same context repeatedly, so that the context elicits the behavior.

SUMMARY:
This 12-week trial will test the efficacy of a personalized, multi-component, personalized text-message delivered behavior change technique (BCT) intervention to encourage habitual hourly physical activity among care providers of persons with Alzheimer's Disease and Alzheimer's Disease Related Dementias (AD/ADRD) via the key mechanism of behavior change (MoBC) of automaticity.

The main question it aims to answer is whether a multi-component, personalized BCT intervention to increase habitual walking of >250 steps/hour will lead to successful development of habitual hourly walking among 50% of caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a caregiver (formal/paid or informal/unpaid) for persons with Alzheimer's Disease or Alzheimer's Disease Related Dementias (AD/ADRD)
* Age >=18 and <=85
* Speak English or Spanish as primary language
* Self-report low levels of physical activity or walking

Exclusion Criteria:

* Individuals who self-report having been informed by a clinician it is medically or physically unsafe to engage in a walking intervention
* Does not own or cannot regularly access a smartphone capable of receiving text messages or accessing the internet
* Does not own or have access to an email address
* Lives outside the United States

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Binary indicator of habit formation | Baseline to intervention period (12 weeks)
  The primary outcome will be a binary indicator of habit formation. A null hypothesis rate of 30 percent will be used. There will be a comparison of the achieved proportion of habitual walking versus this null level, using a 1-sample binomial test with a 2-sided alpha at 5 percent. For the purposes of this current analysis, it is assumed that 50 percent of the sample will achieve habitual hourly walking following the BCT intervention to encourage habit formation. Rate of habit formation will be summarized using the observed proportion along with a 95 percent confidence interval.

SECONDARY OUTCOMES:
Habit formation association with changes in automaticity | Baseline (first 2 weeks of study) and last 2 weeks of intervention
  Examining whether an hourly walking habit formation will be associated with positive changes in cognitive automaticity using Fisher's exact test (5%, 2-sided). Specifically, for each participant, the difference between average automaticity during the last 2 weeks of intervention and average baseline automaticity will be calculated; a positive change is defined as a difference of greater than zero. The rate of habit formation will be compared between the group of participants whose automaticity increased and the participants whose automaticity did not using a Fisher's exact test. Finally, logistic regression will be utilized to assess the effects of automaticity on development of a daily walking habit, with adjustment for other factors, such caregiver demographic characteristics and factors related to caregiving.
Longitudinal association between automaticity and habitual walking over time | Baseline to intervention period (12 weeks)
  Longitudinal associations between the intervention, automaticity, and habitual walking over time will be examined using univariate logistic regression models. These models will provide preliminary estimates of how automaticity change at a given week will impact habit formation, thus informing how the timing of automaticity change will impact habit. Further, weekly automaticity changes will be explored together in a multivariate Bayesian logistic regression model, which will be trained using iPIPE.238
Heterogeneity of treatment effects for habit formation and on changes in automaticity | Baseline to intervention period (12 weeks)
  To examine the heterogeneity of treatment effects for habit formation and on changes in automaticity, analyses of HTEs across participants will be conducted. This will involve examining the heterogeneity in time to achieving habitual hourly walking due to the BCT intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Goodwin, PhD, Principal Investigator — Northwell Health
Locations (1):
- Institute of Health System Science, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Scientific data generated as a result of this research will be shared broadly via OpenScience: https://cos.io/ or a comparable data registry. There will be no identifiable data posted publicly.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, including the statistical analysis plan, will be made available in addition to the informed consent form following completion of recruitment but prior to publication of any data from the current study. De-identified individual participant data will be made available at time of primary outcome manuscript publication, whichever comes last. Data is anticipated to be available on the Open Science Framework or comparable data registry indefinitely.
Access Criteria: All de-identified study data and supporting information will be stored on the Open Science Framework or comparable data registry, a free web application with no access restrictions.